CLINICAL TRIAL: NCT06808672
Title: Plasma Membrane Antigens As Trigger in Cancer-associated Myositis
Brief Title: Biomarkers of Cancer-Associated Myositis
Acronym: MIOSURFACE
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 419/2019/OSS/AUSLRE
Record Dates: First submitted 2024-03-22; First posted 2025-02-05 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Dermatomyositis
Keywords: Dermatomyositis; Immune Checkpoints; Autoantibodies; Cancer Risk
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Sera samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- DM without cancer: Patients with DM who do not have cancer at diagnosis and in the 3-year follow-up period
- DM with cancer: Patients with DM who have cancer at diagnosis or in the 3-years before or after DM diagnosis
- Healthy controls: Subjects without known cancer, autoimmune diseases and infections

SUMMARY:
The project is about dermatomyositis (DM), an autoimmune disease characterized by inflammation in the skeletal muscles and skin. Patients with DM have an increased risk of cancer, with a cancer incidence between 5.5% and 42%. Cancers in these patients are one of the leading causes of death. Some myositis-specific autoantibodies have been discovered and some of them are associated with cancer development. However, DM patients negative for all the known autoantibodies can also develop cancer. The Investigator hypothesized that antibodies against plasma membrane antigens and soluble immune checkpoints can be responsible for the association between cancers and autoimmunity. Therefore, the present study aimed to identify novel antigens and immunological pathways in patients with DM with cancer versus patients with DM without cancer, to identify those patients who need cancer screening. The Investigators focus on soluble immune checkpoint molecules and autoantibodies directed against plasma membrane antigens.

DETAILED DESCRIPTION:
Several studies have reported an association between cancers and autoimmune diseases. Mechanisms underlying this association are largely unknown, but similarity between antigens expressed by cells in tissues targeted by autoimmune reactions and cancer cells is likely one of the drivers. Moreover, chronic inflammation can favor cancer onset.

Among autoimmune diseases, dermatomyositis (DM) has the highest association with cancers. About 25% of patients with DM, over 40 years old, have cancer at the time of diagnosis or develop cancer later. Common cancers include lung, breast, colon, prostate, and ovarian cancers. DM is a systemic inflammatory disease affecting skeletal muscle, skin, and other organs (e.g., lung). Cancer risk in patients with DM is higher compared to age- and sex-matched populations, both before diagnosis and in the three years following diagnosis (standardized incidence ratio: 3.8 - 17.29).

DM is characterized by autoantibodies. Autoantibodies against transcriptional intermediary factor TIF1-gamma, nuclear matrix protein (NXP2), and SUMO1 activating enzyme (SAE1) are detected more frequently in patients with paraneoplastic DM compared to patients without cancers and healthy controls. In contrast, autoantibodies against Jo-1 are detected less frequently. However, the identification of patients with increased cancer risk remains incomplete since DM patients negative for all known autoantibodies also have an increased risk. While TIF1-gamma, NXP2, and Jo-1 are intracellular antigens, plasma membrane antigens are more likely involved in cancer-associated DM due to their accessibility to antibodies.

Immune checkpoint molecules have emerged as key regulators of the immune system, crucial for self-tolerance and immune activation. They mainly act as ligand-receptor pairs, but several undergo alternative splicing, generating soluble isoforms. The production of soluble forms of immune checkpoints in DM is scarcely known.

Autoantibodies against extracellular antigens and soluble immune checkpoints may contribute to the association between cancers and autoimmunity. Identifying circulating markers deregulated in cancer-associated DM will enable the identification of patients at risk, facilitating timely screening and interventions.

Patients with dermatomyositis (DM) have an increased risk of developing tumors, making early detection crucial due to their worse prognosis. The currently known autoantibodies, such as anti-TIF1-gamma, anti-NXP2, and anti-SAE1, fail to identify all DM patients with associated tumors. Additionally, about 35% of DM patients are negative in standard autoantibody screenings but still exhibit a higher tumor risk. So far, the identified autoantibodies in cancer-associated DM target intracellular antigens, which are unlikely to have a direct pathogenic role as they cannot bind their targets under physiological conditions. Soluble immune checkpoints are believed to mediate the relationship between DM and cancer, potentially serving as biomarkers. The study hypothesizes that autoantibodies against cell surface antigens, which are more likely to be pathogenic, may be present in tumor-associated DM. It also proposes that changes in soluble immune checkpoint levels might contribute to DM-associated tumor development and could help identify at-risk patients.

This is a prospective and retrospective study. For the prospective part, serum samples will be collected at the time of enrollment, before the initiation of chemotherapy or immunotherapy. For the retrospective part, patients enrolled in the study must have an available serum sample stored at -80°C, and potentially a muscle biopsy, fixed in formalin and embedded in paraffin, taken during the diagnostic phase.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years.
* Diagnosis of DM.
* Informed Consent

Exclusion Criteria:

* Chemotherapy at the time of the peripheral venous blood draw.
* Therapy with biologic drugs at the time of the peripheral venous blood draw.
* Necrotizing autoimmune myopathy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with DM during rheumatologic visits of the national health system
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of autoantibodies against surface proteins in patients with dermatomyositis (DM) with and without cancer. | At enrollement
  Serum samples from patients with DM with and without cancer will be tested for their ability to bind various cell lines surface antigens through immunofluorescence assays on live cells. Median fluorescence intensity will be evaluated. These analyses will determine whether there are differences in the levels of autoantibodies between the serum samples from patients with and without cancer. Potential autoantigens will be identified by immunoprecipitation of cell lysates with sera followed by mass spectrometry.
Identification of soluble immune checkpoint molecules in patients with dermatomyositis (DM) with and without cancer. | At Enrollment
  Levels of 14 soluble immune checkpoint molecules will be quantified in serum samples using the Magpix technology (ProcartaPlex Immuno-Oncology Checkpoint Panel 1). The target molecules include: BTLA, GITR, HVEM, IDO, LAG-3, PD-1, PD-L1, PD-L2, TIM-3, CD28, CD80, CD137, CD27, and CD152. Concentrations of soluble immune checkpoints will be evaluated. These analyses will determine whether there are differences in the levels of these molecules between the serum samples from patients with and without cancer.

SECONDARY OUTCOMES:
Expression of autoantigens in muscle biopsy samples from DM patients and cancer samples | At Enrollment
  The expression of novel autoantigens will be tested using the immunohistochemistry technique in muscle biopsy samples from dermatomyositis (DM) patients, as well as in samples from ovarian, breast, and colon carcinomas, and normal tissues. Differences in the expression pattern of autoantigens between the DM patient samples and tumor samples will be identified
Expression of autoantibodies against surface proteins in patients with dermatomyositis (DM) compared to healthy controls. | At Enrollment
  Median fluorescence intensities obtained after incubation of live cells with sera from DM patients will be compared to those obtained with sera from healthy subjects. These measurements will determine whether there are differences in the levels of these molecules between the serum samples from DM patients and healthy subjects.
Expression of soluble immune checkpoint molecules in patients with dermatomyositis (DM) compared to healthy controls. | At Enrollment
  The levels of 14 soluble immune checkpoint molecules will be compared between serum samples from DM patients and healthy subjects. These measurements will determine whether there are differences in the levels of these molecules between the serum samples from DM patients and healthy subjects.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Universitaria Consorziale Policlinico di Bari, Bari
  - AUSL-IRCCS di Reggio Emilia, Reggio Emilia

IPD SHARING:
Plan to Share IPD: No